CLINICAL TRIAL: NCT05502276
Title: Endoscopic Full Thickness Resection (EFTR) Versus Endoscopic Submucosal Dissection (ESD) in the Treatment of Difficult Colorectal Lesions With Dimensional Cut-off ≤ 30mm: Laterally Spreading Tumor Non Granular Type (LST-NG), "no Lift" Lesions and Residual / Relapses of Previous Resections. Endoscopic.
Brief Title: Full Thickness Resection or Endoscopic Submucosal Dissection for Difficult Colorectal Lesions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giulio Antonelli, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESECT
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Submucosal Dissection (ESD) (Active Comparator): The Endoscopic Submucosal Dissection (ESD) procedures will be performed with the devices commonly used at the Services of Endoscopy of the Centers participating in the study. There are several models of knives on the market, produced by different companies, all considered equally effective by international guidelines.
  Interventions: Procedure: Endoscopic Submucosal Dissection (ESD)
- Endoscopic Full-Thickness Resection (EFTR) (Experimental): The FTRD® (Full Thickness Resection Device; Ovesco Endoscopy, Tübingen, Germany) is the only over-the-scope device designed to undergo Endoscopic Full-Thickness Resection (EFTR) using a "clip-and-cut" technique. It consists of a 14 mm modified over-the-scope-clip (OTSC) mounted on the outside of a 23 mm cap, which has a preloaded 13 mm monofilament loop at the end. This device received the CE mark for the lower digestive tract in September 2014 and its efficacy and safety have been evaluated in preclinical studies and clinical trials.
  Interventions: Procedure: Endoscopic Full-Thickness Resection (EFTR)

INTERVENTIONS:
Procedure: Endoscopic Full-Thickness Resection (EFTR) — Full Thickness Endoscopic Resection using the FTRD Ovesco Device
  Arms: Endoscopic Full-Thickness Resection (EFTR)
Procedure: Endoscopic Submucosal Dissection (ESD) — Standard Endoscopic Submucosal Dissection using standard procedure described in international guidelines.
  Arms: Endoscopic Submucosal Dissection (ESD)

SUMMARY:
Compare the efficacy and safety of endoscopic resection a full thickness (EFTR) with Full Thickness Resection Device (FTRD) System versus endoscopic submucosal dissection (ESD) in the treatment of Laterally Spreading Tumor Non Granular Type (LST-NG), "no lift" lesions colon and residual / relapse on scars from previous resections endoscopic colon. The dimensional cut off of these lesions is ≤30mm

ELIGIBILITY:
Inclusion criteria:

* patients of age >18 years
* Laterally Spreading Tumor Non Granular Type (LST-NG) ≤ 3cm in diameter
* "no-lift" colic injuries ≤ 3cm in diameter
* residual / recurrence on the scar of previous endoscopic resections of the colon ≤ 3cm in diameter

Exclusion criteria:

* pregnant women
* failure to accept or understand the consent to participate in the study
* patients with severe coagulopathies
* patients with short life expectancy (Charlson comorbidity index ≥8)
* patients with expired general clinical conditions (American Society of Anesthesiologists score ≥3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
En-bloc resection rate | 1 year
  the rate of one-piece resection of the lesions
R0 resection rate | 1 year
  percentage of patients with histologically negative lateral and deep margins

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Dei Castelli, Ariccia, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andrisani G, Hassan C, Pizzicannella M, Pugliese F, Mutignani M, Campanale C, Valerii G, Barbera C, Antonelli G, Di Matteo FM. Endoscopic full-thickness resection versus endoscopic submucosal dissection for challenging colorectal lesions: a randomized trial. Gastrointest Endosc. 2023 Dec;98(6):987-997.e1. doi: 10.1016/j.gie.2023.06.009. Epub 2023 Jun 28. PMID 37390864